CLINICAL TRIAL: NCT02410148
Title: Non-invasive Absolute Intracranial Pressure (ICP) Measurement in Patients With Open-angle Glaucoma and Papilledema
Brief Title: aICP in Glaucoma and Papilledema
Acronym: aICP Ophtha
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, PD Dr.med. HE Killer, Professor, Kantonsspital Aarau
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: aICP Ophtha
Record Dates: First submitted 2015-03-23; First posted 2015-04-07 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Open-angle Glaucoma; Papilledema
Keywords: open-angle glaucoma; papilledema; non-invasive ICP; Intracranial pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Papilledema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Papilledema (Active Comparator): non-invasive aICP measurement in patientes with papilledema
  Interventions: Device: Non-invasive ICP measurement (Vittamed 305)
- open angle glaucoma (Active Comparator): non-invasive aICP measurement in patients with glaucoma
  Interventions: Device: Non-invasive ICP measurement (Vittamed 305)

INTERVENTIONS:
Device: Non-invasive ICP measurement (Vittamed 305) — The non-invasive method is based on two-depth TCD technique for simultaneously measuring flow velocities in the intracranial and extracranial segments of the ophthalmic artery (OA).

SUMMARY:
Glaucoma remains a disease with an unclear and complex underlying pathophysiology. Recently, researchers have emphasized not only intraocular pressure (IOP) or vascular dysregulation, but also translaminar pressure's (TPG) role in glaucoma (TPG=IOP-ICP). A higher TPG may lead to abnormal function and optic nerve damage due to changes in axonal transportation, deformation of the lamina cribrosa, altered blood flow, or a combination thereof leading to glaucomatous damage. However only invasive ICP measurements are available within the contemporary medicine. The ideas for non-invasive ICP measurement have been approached since about 1980. Most of the proposed technologies were based on ultrasound and were capable of monitoring blood flow in intracranial or intraocular vessels, cranium diameter, or acoustic properties of the cranium. Broad research has extended into sonography of optic nerve sheath and its relation with elevated ICP. However, most of these correlation-based methods had the same problem-the need of individual patient specific calibration. Seeking to measure absolute ICP values, researchers from Kaunas University of Technology created a non-invasive method, which does not need a patient specific calibration. The method is based on direct comparison of ICP value with the value of pressure Pe that is externally applied to the tissues surrounding the eyeball. Intracranial segment of ophthalmic artery (OA) is used as a natural sensor of ICP and extracranial segment of OA is used as a sensor of Pe. The special two depth transcranial Doppler (TCD) device is used as a pressure balance indicator when ICP = Pe.

The aim of our study is to assess TPG in patients with primary open open-angle glaucoma (POAG). In addition the investigators want to measure ICP in patients with papilledema (PE) in order to compare them with glaucoma patients.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy leading to the retinal ganglion cell death and typical optic nerve head (ONH) damage [1]. It remains a disease with an unclear and complex underlying pathophysiology. Intraocular pressure (IOP) is the main and only modifiable risk factor for glaucoma [2]. Although lowering IOP helps to decelerate or stabilize the disease, a vast number of patients still show signs of glaucoma despite an IOP within normal range. Clearly other pathogenetic mechanisms beyond IOP are involved in the pathogenesis of glaucoma for certain individuals. Non-IOP factors such as lower systolic ocular perfusion pressure (OPP), reduced ocular blood flow, cardiovascular disease, and low systolic blood pressure (BP) have been identified as risk factors for primary open-open-angle glaucoma (POAG) [3-6]. Evidence shows that non-IOP factors can impact the apoptotic process associated with glaucoma [7].

Recently, researchers have emphasized not only IOP or vascular dysregulation, but also intracranial pressure's (ICP) role in glaucoma [8-10]. The optic nerve is exposed not only to IOP in the eye, but also to ICP as it is surrounded by cerebrospinal fluid (CSF) in the subarachnoid space. Because the lamina cribrosa separates these two pressurized regions [11], the decrease in pressure that occurs across the lamina cribrosa (IOP-ICP) is known as the translaminar pressure gradient (TPG). A higher TPG may lead to abnormal function and optic nerve damage due to changes in axonal transportation, deformation of the lamina cribrosa, altered blood flow, or a combination thereof leading to glaucomatous damage. Besides, TPG may be the primarily pressure-related parameter for glaucoma [12-15], since the ONH is located at the junction between the intraocular space and the orbital retrobulbar space.

However, the role of TPG still remains unknown, because only invasive ICP measurements are available within the contemporary medicine (lumbar puncture or punction of brain ventricles-for patients with severe brain injury). The ideas for noninvasive ICP measurement have been appearing since about 1980. Numerous methods for finding the objects or physiological characteristics of cerebrospinal system that would be related to the ICP and its monitoring have been sought by many authors. Most of the proposed technologies were based on ultrasound and were capable of monitoring blood flow in intracranial or intraocular vessels, cranium diameter, or acoustic properties of the cranium [16]. Broad research has extended into sonography of optic nerve sheath and its relation with elevated ICP [17]. However, most of these correlation-based methods had the same problem-the need of individual patient specific calibration. Seeking to measure absolute ICP values, researchers from Kaunas University of Technology created a noninvasive method, which does not need a patient specific calibration [18, 19]. The method is based on direct comparison of ICP value with the value of pressure Pe that is externally applied to the tissues surrounding the eyeball. Intracranial segment of ophthalmic artery (OA) is used as a natural sensor of ICP and extracranial segment of OA is used as a sensor of Pe. A special two depth transcranial Doppler (TCD) device [18, 19] is used as a pressure balance indicator when ICP = Pe. Accuracy, precision, sensitivity, specificity, and diagnostic value of this method were proven with healthy subjects and patients with neurological diseases. This device has not yet been used in clinical studies to investigate TPG significance in glaucoma. The aim of our study is to assess TPG in patients with primary open open-angle glaucoma (POAG). In addition the investigators want to measure ICP in patients with papilledema (PE) in order to compare them with glaucoma patients.

The non-invasive ICP measurement using two deeps TCD device allows us to get ICP values from immediate vicinity of optic nerve, which in turn very important in term of understanding the pathophysiology of such conditions like PE and POAG.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed POAG or PE
* Age: ≥18 years at admission
* Informed consent

Exclusion Criteria:

* Patients with wounds, scars including the front orbital region.
* Intraocular pressure range bellow 12 or above 25 mmHg

  > As the aim of the study is to analyze the role of TPG in the progression of POAG and PE, the study focusses on patients with normal IOP (12-25 mmHg)
* Patients with any known ocular condition that - according to an Ophthalmologist - may be worsened by sustained eye pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-07 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
TPG (Translaminar Pressure Gradiant) | Day 1
  TPG= (IOP-ICP)

SECONDARY OUTCOMES:
Arterial blood pressure | Day 1
MD (Mean Deviation) in Visual Field | Day 1
Average RNFL (retinal nerve fiber layer) thickness | Day 1
BCVA (best corrected visual acuity) | Day 1
Adverse Events | Day 14 (+/- 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hanspeter Killer, MD, Principal Investigator — Department of Ophthalmology, Kantonsspital Aarau, Aarau, Switzerland
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland